CLINICAL TRIAL: NCT06278142
Title: Development of a Web-Based Self-Help System for Reducing Procrastination Based on Cognitive Behavioural Approach: Procrastinate
Brief Title: Web-Based Cognitive Behavior Therapy for Procrastination
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Anadolu University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ERTELEME_1
Record Dates: First submitted 2024-02-19; First posted 2024-02-26 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Mental Health Issue
Keywords: Web-based intervention; Cognitive Behavioral Therapy; Procrastination
MeSH Terms: interventions — Counseling

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Guided Web-Based Intervention (Experimental): Participants in this group will use the web-based intervention with guidance support.
  Interventions: Other: Internet Based Intervention - GUIDED
- Without Guidance Web-Based Intervention (Experimental): Participants in this group will use the web-based intervention without guidance support.
  Interventions: Other: Internet Based Intervention - WİTHOUT GUİDANCE
- Waitlist (No Intervention): Participants will have no contact with the study team during the waiting period.

INTERVENTIONS:
Other: Internet Based Intervention - GUIDED — In the expert-supported application, each participant will be sent a folder to be shared by the user and the guide via Google Drive, and the user is expected to perform the application in the folder. A module is added to the folder every Monday and the participant is asked to complete the relevant module until Friday of the same week. In the following two days, a feedback message is provided by the expert, taking into account the user's responses.
  Arms: Guided Web-Based Intervention
Other: Internet Based Intervention - WİTHOUT GUİDANCE — The developed implementation plan is communicated to the participants without expert support and their participation is ensured. A common folder will be created with the participants accepted to the study and in the group without expert support, and the process is managed by transmitting the module to the user via the folder every Monday.
  Arms: Without Guidance Web-Based Intervention

SUMMARY:
The main purpose of this study is to present the development process and project flow of an internet-based self-help intervention programme to reduce the level of procrastination among university students.

DETAILED DESCRIPTION:
In the process of developing the intervention programme, a literature review on procrastination was review on procrastination and it was found that procrastination is a problem for university students in Turkey and the need for an effective intervention programme was identified intervention programme. The existing evidence on the effectiveness of web-based The existing evidence on the effectiveness of web-based intervention programmes was reviewed in the literature developed to address procrastination. In Turkey, web-based interventions are one of the new areas of research. There is no web-based study on procrastination in the Turkish literature. The ERTELE-ME intervention is an internet-based intervention programme consisting of five modules. The intervention programme is deliveredin a guided or self-guided format. The Google Drive service will be used to deliver themodules to the participants.

ELIGIBILITY:
Inclusion Criteria:

* volunteering to participate in the study
* being 18 years of age or older
* being an undergraduate student
* having internet access and an e-mail address with gmail extension
* getting a score above 3.5 points from the Tuckman Procrastination Behaviour Scale, having a score lower than 20 points for the depression sub-dimension, 15 points for the anxiety sub-dimension and 19 points for the stress sub-dimension of the DASS 21 scale (the participant is expected to meet all sub-dimension conditions).

Exclusion Criteria:

* not being in a psychological help process
* not having any psychiatric diagnosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2024-03 (Estimated); Primary Completion 2024-04 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Tuckman Procrastination Behaviour Scale | Time Frame: Pre-test, post-test (5 weeks later from pre-test), follow up (10 weeks later from pre-test)
  Turkish adaptation of the scale consists of 14 items, five-point Likert type (1: strongly disagree-5: strongly agree) and one dimension. The evaluation of the Tuckman Procrastination Behaviour scale is made by taking the average of all items. The maximum score that can be obtained from the scale is expressed as five and the minimum score as one.
Cognitive Distortions Questionnaire | Time Frame: Pre-test, post-test (5 weeks later from pre-test), follow up (10 weeks later from pre-test)
  Turkish adaptation of the form was developed by Batmaz et al. (2015) and consists of 15 items of 9 Likert type. The scale items can be used in short and ultra short form.The 9-item short form will be used to collect data from the study group. The 9-item short form will be used to collect data from the study group.
Time Management Scale | Time Frame: Pre-test, post-test (5 weeks later from pre-test), follow up (10 weeks later from pre-test)
  The lowest score that can be obtained from the scale is 27 and the highest score is 135 (Alay & Koçak, 2002). It was deemed appropriate for the evaluation of time management skills in the study group.
Attitude Scale for Internet-Based Interventions | Time Frame: Pre-test, post-test (5 weeks later from pre-test), follow up (10 weeks later from pre-test)
  Apolinário-Hagen et al. (2018) is a measurement tool consisting of 16 items adapted into Turkish by Özer et al. (in the publication stage). Scale consists of two sub-dimensions named as "Perceived Usefulness and Usefulness" and "Relative Advantage and Comparability".

SECONDARY OUTCOMES:
Depression Anxiety Stress Scale-21 (DASS-21) | Time Frame: Pre-test, post-test (5 weeks later from pre-test), follow up (10 weeks later from pre-test)
  Depression Anxiety Stress Scale (DASS-21) is used to assess depression, stress and anxiety levels.

OTHER OUTCOMES:
Sociodemographic Information Form | [Time Frame: Pre-test]
  This form will assess age, gender and whether the participant has received psychotherapy/counselling or medication before as potential covariates.